CLINICAL TRIAL: NCT05418543
Title: Contrast-enhanced Endoscopic Ultrasound in Diagnosis of Inoperable Bile Duct Tumors
Brief Title: CH-EUS in Diagnosis of Inoperable Bile Duct Tumors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Institutul Regional de Gastroenterologie & Hepatologie Prof. dr. Octavian Fodor (Other)
Responsible Party: Principal Investigator, Rares-Ilie Orzan, Doctor, Institutul Regional de Gastroenterologie & Hepatologie Prof. dr. Octavian Fodor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 1509/03.02.2022
Record Dates: First submitted 2022-06-07; First posted 2022-06-14 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Inoperable Disease; Bile Duct Cancer
MeSH Terms: conditions — Bile Duct Neoplasms | interventions — Biopsy, Fine-Needle

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EUS-FNA (Experimental)
  Interventions: Procedure: Endoscopic ultrasound with fine needle biopsy
- CH-EUS-FNA (Experimental)
  Interventions: Procedure: Endoscopic ultrasound with fine needle biopsy

INTERVENTIONS:
Procedure: Endoscopic ultrasound with fine needle biopsy — Patients with unresectable bile duct tumors will be investigated by either CH-EUS with FNA or conventional EUS with FNA

SUMMARY:
VALIDATION OF THE SUPERIORITY OF CONTRAST ENHANCED ENDOSCOPY TO STANDARD ENDOSCOPY IN THE DIAGNOSIS OF BILE DUCT TUMORS

ELIGIBILITY:
Inclusion Criteria:

* Bile duct tumor diagnosed at endoscopic US, CT scan or MRI
* INR<1.5; platelets > 50.000
* written consent form

Exclusion Criteria:

* INR>1.5; platelets < 50.000
* duodenal invasion or stenosis
* patients denial
* previous treatment for hepato-biliary tumors

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
CH-EUS FNA has higher diagnostic accuracy for bile tuct tumors | one week
  To asses if CH-EUS FNB is superior to CH-EUS FNA when assessing bile duct tumors. To determine the diagnostic accuracy, sensitivity and sensibility.

CONTACTS AND LOCATIONS:
Overall Officials: Andrada Seicean, Professor, Study Director — andradaseicean@gmail.com
Locations (1):
- IRGH "O. Fodor", Cluj-Napoca, Cluj, Romania

IPD SHARING:
Plan to Share IPD: No